CLINICAL TRIAL: NCT05667688
Title: A Phase 1b, Open-Label, Parallel Single-Dose Study to Evaluate the Pharmacokinetics and Pharmacodynamics of Tinlarebant in Healthy Volunteers Aged 50-85
Brief Title: Pharmacokinetics and Pharmacodynamics Study of LBS-008 in Healthy Volunteers Aged 50-85
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RBP4 Pty Ltd (Industry)
Collaborators: Belite Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LBS-008-CT06
Record Dates: First submitted 2022-11-15; First posted 2022-12-28 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteer; Dry Age-related Macular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: 5 mg, fasted (Active Comparator): A single dose (5 mg) of tinlarebant will be administered to each study participant on study Day 1.
  Interventions: Drug: Tinlarebant (LBS-008)
- Cohort 2: 10 mg, fasted (Active Comparator): A single dose (10 mg) of tinlarebant will be administered to each study participant on study Day 1.
  Interventions: Drug: Tinlarebant (LBS-008)

INTERVENTIONS:
Drug: Tinlarebant (LBS-008) — A single dose of Tinlarebant (LBS-008) will be administered to each study participant on study Day 1.

SUMMARY:
This is a Phase 1b, parallel single-dose study to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of Tinlarebant when administered as an oral dose to elderly healthy volunteers. This study will evaluate 2 dose levels in 2 cohorts comprising up to a total of 16 participants (8 per cohort). Dose levels will be evaluated in parallel.

DETAILED DESCRIPTION:
This is a Phase 1b, parallel single-dose study to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of tinlarebant when administered as an oral dose to healthy volunteers aged 50-85. Tinlarebant (previously called LBS-008) is being developed as an oral treatment to slow or halt the progression of dry age-related macular degeneration (AMD) and juvenile onset macular degeneration, known as Stargardt disease (STGD). Accumulation of lipofuscin bisretinoids in the retina is associated with several retinal degenerative diseases including dry AMD and STGD. A total of up to 16 healthy volunteers aged 50-85 are planned to be enrolled into 2 cohorts (8 participants per cohort). Participants will receive a single oral dose of tinlarebant, either 5 mg (Cohort 1) or 10 mg (Cohort 2). The total maximum study duration for participants in this study is 45 days, inclusive of visit windows. This includes a screening period of up to 27 days (Day -28 to Day -2), confinement to the clinical facility over 2 nights (Day -1 to Day 2) and 5 outpatient visits including the EOS visit or Day 15. Tinlarebant will be administered in tablet form; a single tinlarebant tablet will contain 5 mg of IP. Participants in Cohort 1 will receive 1 tinlarebant tablet (5 mg dose) and participants in Cohort 2 will receive 2 tinlarebant tablets (10 mg dose). Enrolment and dosing of participants in Cohorts 1 and 2 may occur concurrently. Healthy volunteers aged 50-85, will be screened between Day -28 and Day -2, inclusive. Participants will be admitted to the clinical facility on Day -1 with tinlarebant dosing to occur on the following day (Day 1). All participants will be dosed under fasted conditions. Participants will be confined at the clinical facility from Day -1 through to Day 2 with discharge following completion of all PK and PD blood sample collections and other scheduled assessments on Day2. If participants experience any clinically significant (CS) AEs during the confinement period, they may remain in the clinical facility for further observation at the discretion of the Principal Investigator (PI). Blood samples for PK and PD analysis will be collected pre-dose and at timepoints up to 24 hours (Day 2) post-dose during the confinement period. Participants will be required to attend the clinic as outpatients on Days 3, 4, 6 and 8 for further safety assessments, PK and PD blood sampling. Participants will then return to the clinical facility for final safety assessments at an end of study (EOS) vision Day 15.

In the event of early study termination prior to the EOS visit (Day 15), participants will be requested to attend the clinic for an early termination (ET) visit.

ELIGIBILITY:
Key inclusion criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Healthy adult male or female, or adult male or female with a stable chronic disease or condition aged 50-85 years of age, inclusive. Adults with stable chronic disease or condition includes adults with no new diagnosis, hospitalisation or changes in medication in the 3 months prior to first dose of study drug on Day 1. Ongoing concomitant medications associated with the stable disease or condition, including over-the-counter (OTC) medications and herbal/vitamin supplements taken by volunteers, will be recorded and reviewed by the PI (or delegate) to determine whether the volunteer is suitable for inclusion in the study. In conducting this review, the PI (or delegate) must consider Exclusion Criteria 11, 12, 13 and 14.
3. The volunteer is considered by the Investigator to be in stable health

Key exclusion criteria :

1. Presence of CS cardiovascular, pulmonary, hepatic, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease, or any other condition that, in the opinion of the Investigator, would jeopardise the safety of the participant or the validity of the study results.
2. Had a CS new illness within 1 month prior to the screening visit, with the exception of fully resolved gastrointestinal illness at least 14 days prior to the screening visit, fully resolved minor colds (e.g., only cold and flu-like symptoms) that occurred within 1 month prior to the screening visit, and fully resolved corona virus disease 2019 (COVID-19) infections if resolved at least 14 days prior to the screening visit and 30 days prior to confinement to the clinical facility.
3. A history of uncontrolled hypertension, coronary artery disease, or any other significant cardiovascular disease.
4. A history of uncontrolled diabetes. Volunteers with fully resolved gestational diabetes will be eligible to participate in the study.
5. A history of unexplained loss of consciousness, epilepsy or other seizure disorder, or cerebrovascular disease.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
To measure the pharmacokinetics (PK) of tinlarebant in plasma following a single oral dose in healthy volunteers aged 50-85. | Up to 168 hours
  Area under the plasma concentration versus time curve from time 0 to the last time point with quantifiable concentration (AUC0-t)
To measure the pharmacokinetics (PK) of tinlarebant in plasma following a single oral dose in healthy volunteers aged 50-85. | Up to 168 hours
  Area under the plasma concentration versus time curve from time 0 extrapolated to infinity (AUC0-inf)
To measure the pharmacokinetics (PK) of tinlarebant in plasma following a single oral dose in healthy volunteers aged 50-85. | Up to 168 hours
  Maximum observed plasma concentration (Cmax)
To measure the pharmacokinetics (PK) of tinlarebant in plasma following a single oral dose in healthy volunteers aged 50-85. | Up to 168 hours
  Time of maximum observed plasma concentration (Tmax)
To measure the pharmacokinetics (PK) of tinlarebant in plasma following a single oral dose in healthy volunteers aged 50-85. | Up to 168 hours
  Apparent plasma terminal elimination half-life (t1/2)
To measure the pharmacokinetics (PK) of tinlarebant in plasma following a single oral dose in healthy volunteers aged 50-85. | Up to 168 hours
  Terminal elimination rate constant (λz)
To measure the pharmacokinetics (PK) of tinlarebant in plasma following a single oral dose in healthy volunteers aged 50-85. | Up to 168 hours
  Apparent total body clearance (CL/F)
To measure the pharmacokinetics (PK) of tinlarebant in plasma following a single oral dose in healthy volunteers aged 50-85. | Up to 168 hours
  Apparent volume of distribution (Vz/F)
To measure the concentrations of retinol-binding protein 4 (RBP4), a pharmacodynamic (PD) biomarker, in plasma following a single oral dose in healthy volunteers aged 50-85 | Up to 168 hours
  Time of minimal RPB4 levels post-dose (Tmin)
To measure the concentrations of retinol-binding protein 4 (RBP4), a pharmacodynamic (PD) biomarker, in plasma following a single oral dose in healthy volunteers aged 50-85 | Up to 168 hours
  Maximal suppression to RBP4 expressed as minimum concentration of RBP4 (Cmin)
To measure the concentrations of retinol-binding protein 4 (RBP4), a pharmacodynamic (PD) biomarker, in plasma following a single oral dose in healthy volunteers aged 50-85 | Up to 168 hours
  Maximal suppression to RBP4 expressed as percent (%) of baseline concentration of RBP4 (C%bmin)
To measure the concentrations of retinol-binding protein 4 (RBP4), a pharmacodynamic (PD) biomarker, in plasma following a single oral dose in healthy volunteers aged 50-85 | Up to 168 hours
  Level of RBP4 at 12 hours as concentration (C12h)
To measure the concentrations of retinol-binding protein 4 (RBP4), a pharmacodynamic (PD) biomarker, in plasma following a single oral dose in healthy volunteers aged 50-85 | Up to 168 hours
  Level of RBP4 at 12 hours as percent of baseline concentration (C%b12h)
To measure the concentrations of retinol-binding protein 4 (RBP4), a pharmacodynamic (PD) biomarker, in plasma following a single oral dose in healthy volunteers aged 50-85 | Up to 168 hours
  Level of RBP4 at 24 hours as concentration (C24h)
To measure the concentrations of retinol-binding protein 4 (RBP4), a pharmacodynamic (PD) biomarker, in plasma following a single oral dose in healthy volunteers aged 50-85 | Up to 168 hours
  Level of RBP4 at 24 hours as percent of baseline concentration (C%b24h)
To measure the concentrations of retinol-binding protein 4 (RBP4), a pharmacodynamic (PD) biomarker, in plasma following a single oral dose in healthy volunteers aged 50-85 | Up to 168 hours
  Half-life for recovery of RBP4 to baseline levels (PDt1/2)

SECONDARY OUTCOMES:
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Incidence, type, severity, and relationship of AEs/serious AEs (SAEs), including withdrawals due to AEs;
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in vital sign measurements (systolic and diastolic blood pressure (BP))
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in vital sign measurements (heart rate (HR))
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in vital sign measurements (respiratory rate)
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in vital sign measurements (body temperature)
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in electrocardiogram (ECG) parameters (RR interval)
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in electrocardiogram (ECG) parameters (PR interval)
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in electrocardiogram (ECG) parameters (QRS width)
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in electrocardiogram (ECG) parameters (QT interval)
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in electrocardiogram (ECG) parameters (QTcB)
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in electrocardiogram (ECG) parameters (QTcF)
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in visual acuity scores
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Changes from baseline in colour vision scores
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Ocular examination assessments (slit lamp biomicroscopy)
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Ocular examination assessments (dilated ophthalmoscopy)
To investigate the systemic and ocular safety and tolerability of a single oral dose of tinlarebant in healthy adult volunteers aged 50-85. | Up to 15 days
  Ocular examination assessments (intraocular pressure)

OTHER OUTCOMES:
To measure the concentration of retinol, a PD biomarker , in serum following a single oral dose of tinlarebant in healthy volunteers aged 50-85. | Up to 168 hours
  Serum retinol concentration for each participant will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Sam Francis, Principal Investigator — Nucleus Network - Melbourne
Locations (1):
- Nucleus Network, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No
After completion of the study, data may be considered for reporting at a scientific meeting or for publication in a scientific journal. In these cases, the sponsor will be responsible for these activities and will work with the investigators to determine how the manuscript is written and edited, the number and order of authors, the publication to which it will be submitted, and any other related issues. The sponsor has final approval authority of all such issues. Data are the property of the sponsor and cannot be published without their prior authorization, but data and any publication thereof will not be unduly withheld.